CLINICAL TRIAL: NCT05751668
Title: An Early Phase and Phase II Clinical Trial to Evaluate Ganglioside-Monosialic Acid (GM1) for Preventing Paclitaxel-Associated Neuropathy
Brief Title: Finding an Effective Dose of GM1 to Reduce or Prevent Neuropathy (Numbness or Weakness) Due to Treatment With Paclitaxel (Phase II)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A222101; NCI-2022-04929 (Other: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Chemotherapy-Induced Peripheral Neuropathy; Metastatic Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Taxes; G(M1) Ganglioside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (paclitaxel, GM1) (Experimental): Patients receive GM1 IV 1 hour prior to paclitaxel administration and paclitaxel IV weekly for 12 weeks or 3 weeks on/1 week off for 12 doses.
  Interventions: Drug: Paclitaxel; Drug: Monosialotetrahexosylganglioside; Other: Questionnaire Administration; Other: Quality-of-life assessment
- Arm II (paclitaxel, placebo) (Placebo Comparator): Patients receive placebo IV 1 hour prior to paclitaxel administration and paclitaxel IV weekly for 12 weeks or 3 weeks on/1 week off for 12 doses.
  Interventions: Drug: Paclitaxel; Other: Questionnaire Administration; Other: Quality-of-life assessment; Drug: Placebo Administration

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol
Drug: Monosialotetrahexosylganglioside — Given IV
  Other Names: Ganglioside GM-1; GM-1; GM1; Monosialoanglioside GM1
  Arms: Arm I (paclitaxel, GM1)
Other: Questionnaire Administration — Ancillary Studies
Other: Quality-of-life assessment — Ancillary Studies
Drug: Placebo Administration — Given IV
  Arms: Arm II (paclitaxel, placebo)

SUMMARY:
This phase II trial tests the safety, side effects, and best dose of monosialotetrahexosylganglioside (GM1) and whether it works in reducing or preventing chemotherapy-induced peripheral neuropathy (CIPN) in patients with breast cancer that has spread from where it first started (primary site) to other places in the body (metastatic) who are receiving treatment with paclitaxel. Chemotherapy drugs, such as paclitaxel, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Exposure to chemotherapy drugs like paclitaxel may cause a side effect called CIPN, which is a condition of weakness, numbness, and pain from nerve damage (usually in the hands and feet). GM1 is a part of the body's natural system that insulates nerves and helps to protect nerves from damage. Giving GM1 may help reduce or prevent CIPN in breast cancer patients receiving treatment with paclitaxel.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain data to further support the safety of increasing monosialotetrahexosylganglioside (GM1) doses when given on day 1, concomitantly with paclitaxel. (Early phase) II. To evaluate the preliminary efficacy of GM1 compared with placebo at preventing paclitaxel-induced peripheral neuropathy sensory symptoms as measured by the six individual Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy 20 (QLQ-CIPN20) questions that quantify numbness (N), tingling (T), and pain in the fingers/hands and toes/feet. (Phase II)

SECONDARY OBJECTIVES:

I. To obtain additional data to support the safety of GM1 in the treated population. (Phase II) II. To obtain data to support that GM1 looks promising for preventing/decreasing acute paclitaxel pain syndrome as measured by the Acute Pain Syndrome Questionnaire. (Phase II)

EXPLORATORY OBJECTIVES:

I. Conduct of this clinical trial provides the opportunity to facilitate the better understanding of the natural history of paclitaxel-induced neuropathy, akin to what is being examined in a currently active trial, S1714. (Phase II) II. This clinical trial also provides an opportunity to conduct correlative studies to understand the mechanism of CIPN and/or identify biomarkers of CIPN or GM1 efficacy. (Phase II) III. To obtain efficacy data to assess the impact of GM1 on the anti-tumor activity of paclitaxel as evaluated by progression-free survival and overall survival. (Phase II)

OUTLINE: This is an early phase dose-escalation study of GM1 followed by a phase II study.

EARLY PHASE: Patients receive GM1 intravenously (IV) over 1 hour either once every 7 days, or once every 7 days for 3 doses followed by one week off, prior to paclitaxel administration.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive GM1 IV 1 hour prior to paclitaxel administration and paclitaxel IV weekly for 12 weeks or 3 weeks on/1 week off for 12 doses.

ARM II: Patients receive placebo IV 1 hour prior to paclitaxel administration and paclitaxel IV weekly for 12 weeks or 3 weeks on/1 week off for 12 doses.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of disease: Histologic diagnosis of metastatic breast cancer in women or men
* Prior treatment- No previous exposure to GM1
* Planned administration of paclitaxel, either given weekly, or weekly 3 weeks on/1 week off, to patients with metastatic cancer at a dose of 80 mg/m^2
* No planned treatment with concurrent immunotherapy
* Score of 1 (none) and/or 2 (a little) on the six individual European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire (QLQ)- chemotherapy-induced peripheral neuropathy (CIPN)20 questions that quantify numbness (N), tingling (T), and pain in the fingers/hands and toes/feet (Items #31-36)
* No diagnosis of fibromyalgia
* No history of significant respiratory tract infection and/or infectious diarrhea within 14 days before registration
* No history of stroke or cerebrovascular accident in the past 6 months prior to registration
* No history of diagnosed neurologic or psychiatric disorders, including epilepsy or dementia
* For women of childbearing potential, not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown.

Therefore, for women of childbearing potential, a negative pregnancy test done =< 7 days prior to registration is required. Of note, a female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

* Ability to complete questionnaires by themselves or with assistance
* In order to complete the mandatory patient-completed measures, participants must be able to speak and/or read English and/or Spanish
* Persons with impaired decision making such that they cannot understand the benefits or risks of trial participation, per the judgement of the consenting clinician, will not be eligible
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN
* No planned use of duloxetine
* No planned use of cryotherapy, compression therapy, or cryocompression therapy at study entry

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2032-03-15 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (Early phase) | 6-7 months
  Defined as the highest dose level that induces dose-limiting toxicity in less than one-third of patients (less than 1 out of 3 or less than 2 out of a maximum of 6 new patients).The constellation of adverse events as scored using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, version (v) 5.0 (CTCAE v5.0) will be summarized by reporting the number and percentage of patients. Specifically, the number and severity of all adverse events (overall and by dose-level) will be tabulated and summarized. The grade 3+ adverse events will also be described and summarized in a similar fashion. Further, all adverse events will be listed by system organ class and preferred term.
Composite response (Phase II) | Up to one year
  Reflects sensory paclitaxel-induced peripheral neuropathy symptom severity and onset. Measured using 6 individual Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy 20 (QLQ-CIPN20) questions that quantify numbness (N), tingling (T) and pain in the fingers/hands and toes/feet. Will calculate the highest (worst) N, T, and pain sensory score obtained anytime during paclitaxel exposure. Response is defined as a patient reporting a highest score of =< 2 without discontinuing the study due to sensory paclitaxel-induced peripheral neuropathy. Chi-squared test will be used. Will report the proportion of patients achieving a composite response in each arm as well as the difference in proportions along with the 90% confidence interval. Will report the estimated odds ratio (monosialotetrahexosylganglioside [GM1]/placebo) and the corresponding 90% confidence interval for the true, but unknown odds ratio. Multiple logistic regression will be used to estimate the intervention

SECONDARY OUTCOMES:
Percentage of patients who received full planned dose of paclitaxel | up to 1 year
  Binary endpoint (yes or no). will graphically look at the percentages of patients receiving full planned paclitaxel doses per cycle within each arm. This is an indirect measure of paclitaxel-induced peripheral neuropathy, as most patients who stop receiving full dose paclitaxel do so because of paclitaxel-induced peripheral neuropathy troubles. In addition to graphically displaying the percentage of patients who receive full dose paclitaxel at each cycle, and according to arm, will make a between-arm comparison in terms of changes in the probability of receiving full dose paclitaxel over the 12 cycles of treatment. For latter analysis, the generalized estimating equations approach will be applied, with inference based on the empirical or sandwich variance estimator.
• Sensory subscale of the European Organization of Research and Treatment of Cancer (EORTC) QLQ-CIPN20 | Up to 1 year
  Serially measured. Item scores are totaled and linearly converted to a 0-100 point scale with higher scores representing fewer symptoms or better quality of life. Will use the area under the curve (AUC) to summarize the serially measured sensory subscale scores. Patients will be analyzed in the arms to which they were randomized. In order to adjust for the stratification factors, the AUC will be computed for the two arms based on estimated parameters from a repeated-measures (means) mixed model.
Rate of grade 3+ Adverse Events | Up to 1 year
  The proportion of patients experiencing a grade 3+ adverse events or toxicities will be described for each treatment arm, and will also be compared between the arms using Fisher's exact tests. Additional summaries and test will be performed as needed.
• Serially measured patient-reported outcome that best describes the patients' aches/pains at its worst in the last 24 hours | In the preceding 24 hours
  Within each arm, the mean score at each time point will be plotted longitudinally for the endpoints measuring aches and pains at its worst. The functional form of the relationship between time and each of these three patient-reported acute neuropathy items is not known. Penalized splines, a smoothing technique which does not require strong assumptions concerning the functional form of the pattern of change in the mean response, will be applied to these longitudinal data. In the two-arm setting (GM1 vs placebo) time trends will be incorporated in a non-parametric fashion, thereby allowing the mean response to change in a highly non-linear, but not predetermined, way. The intervention effect will be incorporated in the model in a parametric fashion, thereby allowing a relatively simple, but powerful, test of the intervention effect on changes in the mean response over time.
Serially measured patient-reported outcome that best describes the patients' aches/pains at its least in the last 24 hours | in the preceding 24 hours
  Within each arm, the mean score at each time point will be plotted longitudinally for the endpoints measuring aches and pains at its least. The functional form of the relationship between time and each of these three patient-reported acute neuropathy items is not known. Penalized splines, a smoothing technique which does not require strong assumptions concerning the functional form of the pattern of change in the mean response, will be applied to these longitudinal data. In the two-arm setting (GM1 vs placebo) time trends will be incorporated in a non-parametric fashion, thereby allowing the mean response to change in a highly non-linear, but not predetermined, way. The intervention effect will be incorporated in the model in a parametric fashion, thereby allowing a relatively simple, but powerful, test of the intervention effect on changes in the mean response over time.
• Serially measured patient-reported outcome that best describes the patients' aches/pains on the average in the last 24 hours | in the preceding 24 hours
  Within each arm, the mean score at each time point will be plotted longitudinally for the endpoints measuring aches and pains on average. The functional form of the relationship between time and each of these three patient-reported acute neuropathy items is not known. Penalized splines, a smoothing technique which does not require strong assumptions concerning the functional form of the pattern of change in the mean response, will be applied to these longitudinal data. In the two-arm setting (GM1 vs placebo) time trends will be incorporated in a non-parametric fashion, thereby allowing the mean response to change in a highly non-linear, but not predetermined, way. The intervention effect will be incorporated in the model in a parametric fashion, thereby allowing a relatively simple, but powerful, test of the intervention effect on changes in the mean response over time.

OTHER OUTCOMES:
Progression free survival (PFS) | Up to 4 years after the end of GM1 treatment
  Distributions of PFS times will be estimated using Kaplan-Meier methodology.
Overall survival (OS) | Up to 4 years after the end of GM1 treatment
  Distributions of OS times will be estimated using Kaplan-Meier methodology.
Serially measured total score of the EORTC QLQ-CIPN20 | On day 1 of each dose prior to GM1, monthly after the end of GM1, at 8, 12, 16, 20, and 24 months after last study treatment
  Will use the AUC to summarize the serially measured EORTC QLQ-CIPN20 scores. Patients will be analyzed in the arms to which they were randomized. In order to adjust for the stratification factors, the AUC will be computed for the two arms based on estimated parameters from a repeated-measures (means) mixed model.
Patient-reported severity and interference of numbness or tingling in hands or feet | On day 1 of each dose prior to GM1, monthly after the end of GM1, at 8, 12, 16, 20, and 24 months after last study treatment
  As measured by the Patient Reported Outcomes version CTCAE (PRO-CTCAE). The maximum grade for each of these events will be recorded for each patient and frequency tables will be generated and presented according to treatment arm. The descriptive analysis of the PRO-CTCAE endpoints will be based on the safety population and analyzed according to the treatment actually received.
Serially measured patient-reported aggregate scores | On day 1 of each dose prior to GM1, monthly after the end of GM1, at 8, 12, 16, 20, and 24 months after last study treatment
  Measured by the 11-item Functional Assessment of Cancer Therapy - Gynecologic Oncology Group-Neurotoxicity 4. Will tabulate all available serially measured PROs at each protocol defined time point and within each arm; furthermore, will graphically display the longitudinal PROs over time. Will compare and contrast the descriptive findings between these CIPN-measuring instruments in this trial and in the corresponding longitudinal data obtained in S1714. No inferential statistics will be generated. Further, these descriptive summaries will be used to better understand these instruments.
Serially measured patient-reported total score | On day 1 of each dose prior to GM1, monthly after the end of GM1, at 8, 12, 16, 20, and 24 months after last study treatment
  Measured by the 5-item Patient Reported Outcomes Measurement Information System-Neuropathic Pain Quality scale. Will tabulate all available serially measured PROs at each protocol defined time point and within each arm; furthermore, will graphically display the longitudinal PROs over time. Will compare and contrast the descriptive findings between these CIPN-measuring instruments in this trial and in the corresponding longitudinal data obtained in S1714. No inferential statistics will be generated. Further, these descriptive summaries will be used to better understand these instruments.

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Morton Plant Hospital, Clearwater, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Saint Anthony's Hospital Cancer Care Center, St. Petersburg, Florida
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin